CLINICAL TRIAL: NCT03474120
Title: Prospective Genetic Study in Patients With Ovarian Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Collaborators: National Research Institute for Family Planning, China (Other Government)
Responsible Party: Sponsor
Other Study IDs: Ovarian-Gene
Record Dates: First submitted 2018-02-05; First posted 2018-03-22 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-07

CONDITIONS: Premature Ovarian Failure; Primary Ovarian Insufficiency; Ovarian Dysgenesis; Diminished Ovarian Reserve
Keywords: Genetic causes; etiology; POI; DOR
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect 5 ml whole blood(in EDTA anticoagulant tube) and sign an informed consent form for patients diagnosed with POI/DOR/ovarian dysgenesis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IVF treatment group: Patients treated with IVF. IVF promotion process, ovulation, fertilization, embryo quality, transplantation and final outcome were collected after the treatment cycle was completed.
  Interventions: Procedure: IVF treatment
- No IVF treatment group: the patients who did not have received IVF treatment .Patients were followed up to collect hormone levels, ultrasound results.

INTERVENTIONS:
Procedure: IVF treatment — Relationship between IVF treatment outcome and genotypes in POI//DOR/ovarian dysgenesis patients
  Other Names: No IVF treatment
  Groups: IVF treatment group

SUMMARY:
genetic screening and etiological analysis was conducted on patients with ovarian insufficiency and decline in ovarian reserve. All patients were enrolled in the IVF-treated and non-IVF-treated groups, followed up for long-term treatment outcomes and genomic screening.

DETAILED DESCRIPTION:
The cause of ovarian insufficiency and decline in ovarian reserve are not clear, but most researchers think the probable causes are mainly three aspects: chromosomal abnormalities, genetic factors and autoimmune diseases，But the majority of patients with normal chromosome karyotype analysis. The screening of pathogenic genes in patients with normal karyotype is the focus of current premature ovarian insufficiency(POI) and decline in ovarian reserve(DOR) etiology, to further explain the pathogenesis of patients, improve the diagnosis of those diseases and Clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as "premature ovarian insufficiency", "diminished ovarian reserve", "primary amenorrhea", " ovarian dysgenesis", " repeated implantation failure"

Exclusion Criteria:

* To rule out polycystic ovary syndrome（PCOS）, iatrogenic factors (such as surgery, radiotherapy and chemotherapy, etc.) lead to premature ovarian insufficiency in patients

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who come to the First Affiliated Hospital of Anhui Medical University Reproductive Center and diagnosed as "premature ovarian insufficiency", "diminished ovarian reserve", "primary amenorrhea", " ovarian dysgenesis", " repeated implantation failure"，Understand the content of the project and sign an informed consent form
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2023-01-24 (Estimated); Study Completion 2023-12-24 (Estimated)

PRIMARY OUTCOMES:
Genotype | 1/4/2018-24/12/2020
  Measure the genotype by genome-wide sequencing of exomes(WES) in subjects.

SECONDARY OUTCOMES:
Dimensions of uterus | 1/4/2018-24/12/2020
  Measure the vertical diameter，transverse diameter and anteroposterior diameter of uterus in millimeters
Antral follicle count | 1/4/2018-24/12/2020
  Measure the basic antral follicle count before controlled ovarian hyperstimulation.
Endometrial thickness | 1/4/2018-24/12/2020
  Measure endometrial thickness of subjects in millimeters.
Live birth rate | 1/4/2018-24/12/2020
  Record the live birth rate of offspring in in both groups.
Neonatal weight | 1/4/2018-24/12/2020
  Record the neonatal weight(in kilogram) of offspring in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yunxia Cao, PhD, Study Director — Reproductive Medicine Center, the First Affiliated Hospital of AMU
Locations (1):
- Reproductive Medicine Center, the First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China